CLINICAL TRIAL: NCT04906460
Title: An Open-label Phase 1b/2 Study of WVE-N531 in Patients With Duchenne Muscular Dystrophy
Brief Title: Open-label Study of WVE-N531 in Patients With Duchenne Muscular Dystrophy (FORWARD-53)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVE-N531-001
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- WVE-N531 (Experimental)
  Interventions: Drug: WVE-N531

INTERVENTIONS:
Drug: WVE-N531 — WVE-N531 is an antisense oligonucleotide (ASO)

SUMMARY:
This is a Phase 1b/2 open-label study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and clinical effects of intravenous (IV) WVE-N531 in patients with Duchenne muscular dystrophy (DMD). To participate in the study, patients must have a documented mutation of the DMD gene that is amenable to exon 53 skipping intervention. This study has 3 parts, Part A, Part B, including Part B Extension Arm, and Part C. Part A is completed. Part B is completed. Following completion of Part B, all patients elected to continue to receive study drug in the optional Part B open-label Extension Arm. Part C has been added to the study and will enroll new patients.

DETAILED DESCRIPTION:
Following completion of Part A, eligible patients rolled over into Part B to continue to receive treatment. In addition, new patients were enrolled up to a total of 11 patients in Part B. All patients received WVE-N531 at 10 mg/kg every other week (Q2W) until competent authority approval of a protocol update, when all patients were switched to Q4W dosing. Muscle biopsies were performed following 24 weeks and for new Part B patients (those that did not take part in Part A) following 48 weeks of treatment. Following completion of Part B, all patients elected to continue to receive study drug at Q4W for up to 1 year in an optional Part B Extension Arm.

For this portion of the study, up to 15 new patients will be enrolled into Part C of the study. All patients will undergo an open muscle biopsy, at baseline and following 24 weeks of treatment.

The primary endpoint for Part B is the measurement of dystrophin protein levels. Participants will also be evaluated for safety, tolerability, digital and functional endpoints.

The primary endpoint for Part C is the measurement of dystrophin protein levels. Participants will also be evaluated for safety, tolerability, digital and functional endpoints. Safety monitoring will occur through 10 months after the last dose.

ELIGIBILITY:
Inclusion Criteria:

Part A and Part B:

1. Part A patients may be screened for Part B upon completion of a washout period of ≥18 weeks from last dose in Part A. New patients may also be screened for Part B
2. Diagnosis of DMD based on clinical phenotype.
3. Documented mutation in the DMD gene associated with DMD that is amenable to exon 53 intervention
4. Score of ≥1 on item 1 or 2 of the shoulder component of the Performance of the Upper Limb (PUL) (Part B ).
5. Ambulatory or non-ambulatory male
6. Stable pulmonary and cardiac function, as measured by the following: (Part B):

1. Reproducible percent predicted forced vital capacity (FVC) ≥50%; 2. Left ventricular ejection fraction (LVEF) >55% in patients <10 years of age and >45% in patients ≥10 years of age, as measured (and documented) by echocardiogram (ECHO) and/or cardiac magnetic resonance imaging (MRI), within 6 months prior to enrollment into the study.

7.Adequate muscle at Screening to perform open muscle biopsies, preferably deltoid.

8. Currently on a stable corticosteroid therapy regimen, defined as initiation of systemic corticosteroid therapy that occurred ≥6 months prior to Screening and no changes in dose ≤3 months prior to Screening visit (Part B ).

Part C

1. New patients to be screened for Part C.
2. Diagnosis of DMD based on clinical phenotype.
3. Documented mutation in the DMD gene associated with DMD that is amenable to exon 53 intervention
4. Score of ≥1 on item 1 or 2 of the shoulder component of the Performance of the Upper Limb (PUL) .
5. Ambulatory male
6. Stable pulmonary and cardiac function, as measured by the following:

1. Reproducible percent predicted forced vital capacity (FVC) ≥50%; 2. Left ventricular ejection fraction (LVEF) >55% in patients as measured (and documented) by echocardiogram (ECHO) and/or cardiac magnetic resonance imaging (MRI), within 6 months prior to enrollment into the study.

7. Adequate muscle at Screening to perform open muscle biopsies, preferably deltoid.

8. Currently on a stable corticosteroid therapy regimen, defined as initiation of systemic corticosteroid therapy that occurred ≥6 months prior to Screening and no changes in dose ≤3 months prior to Screening visit .

Exclusion Criteria:

1. Clinically significant medical finding on the physical examination other than DMD that, in the judgment of the Investigator, will make the patient unsuitable for participation in, and/or completion of the study procedures.
2. Part B and Part C: Major surgery within 3 months prior to Day 1 or planned major surgery for any time during the study.
3. Part B: Diagnosis of active alcohol, cannabinoid, or other substance use disorder (except nicotine) within 6 months prior to the Screening visit
4. Part C: Any recreational substance use (including prescribed cannabinoids), with the exception of nicotine, irrespective of legality, within 2 months prior to Screening and/or unwilling to refrain from such use for the duration of the study.

Ages: 4 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety: Proportion of patients with adverse events (AEs) | Day 1 (initial dose) up to 24 weeks after the last dose of Part A
Part B: Pharmacodynamics: Dystrophin level (% normal dystrophin) as assessed by Western blot of muscle tissue following multiple doses of WVE-N531 | At Week 26 and at Week 50 of Part B
Part C: Pharmacodynamics: Change from baseline dystrophin level (% normal dystrophin) as assessed by a validated assay analysis in muscle tissue following multiple doses of WVE-N531 | At Baseline and following 24 weeks of treatment in Part C

SECONDARY OUTCOMES:
Part A: Pharmacokinetics: Concentration of WVE-N531 in muscle tissue | Day 1 (initial dose) through 2 weeks after the last dose of Part A
Part A: Pharmacodynamics: Dystrophin level (% normal dystrophin) as assessed by Western blot of muscle tissue following multiple doses of WVE-N531 | Day 1 (initial dose) through 2 weeks after the last dose of Part A
Part B: North Star Ambulatory Assessment (NSAA) (Version 2.0), including time to stand and a timed 10-meter walk/run, with a range of 0 to 34 where higher scores indicate better outcome. | Collected at baseline, Weeks 24 and 48 of Part B, at baseline and Weeks 26 and 50 of the Extension Arm
Part B: Performance of the Upper Limb (PUL) (Version 2.0) with a range of 0 to 64 where higher scores indicate a better outcome. | Collected at baseline, Weeks 24 and 48 of Part B, at baseline and Weeks 26 and 50 of the Extension Arm
Part B: Stride Velocity 95th Centile (SV95C)/upper limb outcome (non-ambulatory patients) | Collected at baseline, Weeks 24 and 48 of Part B, at baseline and Weeks 26 and 50 of the Extension Arm
Part C: North Star Ambulatory Assessment (NSAA) (Version 2.0), including time to stand and a timed 10-meter walk/run, with a range of 0 to 34 where higher scores indicate better outcome. | Collected at baseline and Week 24 of Part C
Part C: Performance of the Upper Limb (PUL) (Version 2.0) with a range of 0 to 64 where higher scores indicate a better outcome. | Collected at baseline and Week 24 of Part C
Part C: Stride Velocity 95th Centile (SV95C)/upper limb outcome (non-ambulatory patients) | Collected at baseline and Week 24 of Part C

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (5):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rare Disease Research LLC, Atlanta, Georgia
- Jordan (2):
  - Istiklal Hospital/ Clinical Research Unit, Amman
  - The Specialty Hospital (TSH)/ Advanced Clinical Center, Amman
- Oxford Children's Hospital, Oxford University Hospitals NHS Foundation Trust, Headington, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No